CLINICAL TRIAL: NCT00620633
Title: A Phase I Dose Escalation Trial of WT1-Sensitized T Cells for Residual or Relapsed Leukemia After Allogeneic Hematopoietic Progenitor Cell Transplantation
Brief Title: Dose Escalation Trial of WT1-Sensitized T Cells for Residual or Relapsed Leukemia After Allogeneic Hematopoietic Progenitor Cell Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Atara Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-055
Record Dates: First submitted 2008-02-11; First posted 2008-02-21 (Estimated); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Leukemia; Myelodysplastic Syndrome
Keywords: Bone Marrow
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes

ARMS (1):
- 1 (Experimental): Patients with leukemia or myelodysplastic syndrome (MDS) who, following an HLA-matched allogeneic hematopoietic cell transplant, have relapsed with leukemia as demonstrated morphologically on peripheral blood smear or bone marrow aspirate
  Interventions: Biological: WT1-sensitized T cells

INTERVENTIONS:
Biological: WT1-sensitized T cells — Eligible patients who consent to enter this trial and for whom WT1 sensitized T cells have been generated in vitro, will receive a single dose of allogeneic WT1-sensitized T cells by bolus intravenous infusion. In this phase I trial, 6 dose levels of T cells will be evaluated, in sequential groups of 3 patients. Dose Escalation will be based on the incidence and severity of toxicities.

SUMMARY:
This study will test the safety of giving you specialized white cells from your donor. They are called WT1 sensitized T cells. They have been grown in the lab and are immunized against a protein. The protein is called the Wilms' tumor protein, or WT1. Your leukemic cells make too much of this protein. We want to learn whether the WT1 sensitized T cells will attack the protein and kill the leukemia cells.

ELIGIBILITY:
Inclusion Criteria:

* Prior to receiving treatment, some patients may undergo diagnostic and/or other testing of their WT1 malignancies to determine if their disease is likely to respond to treatment with WT1 specific T cells. Alternatively, blood samples may be required for research tests to ascertain that the WT1-specific T-cells do not contain any cells that could react against the patient. These patients will sign a separate pre-treatment consent. If it is determined that a patient will qualify for and might benefit from infusions of WT1 CTLs, he/she will go on to sign the standard treatment consent for MSKCC IRB # 07-055 and be enrolled and treated on trial, if all other eligibility criteria are met.
* Patients eligible for this trial will include patients with a pathologically confirmed diagnosis of leukemia or myelodysplastic syndrome (MDS) who, following an allogeneic hematopoietic cell transplant, have relapsed with leukemia as demonstrated morphologically on peripheral blood smear or bone marrow aspirate, or have recurrent persistent minimal residual disease as demonstrated by at least 2 sequential testings separated by at least 1 week demonstrating molecular evidence of residual leukemia or MDS by FISH or cytogenetics. In addition, patients who are to receive an allogeneic hematopoietic cell transplant as treatment for a leukemia or myelodysplastic syndrome that has an expected of risk of relapse post transplant of >30% will be eligible to have donor-derived WT1 peptide specific T cells generated prior to or at the time of transplant for immediate use post transplant at such time that the patient is found to have minimal residual disease or relapse. This includes patients with AML or ALL that is either refractory to primary induction therapy or is at any stage later than first relapse for AML or ALL, CML in a secondary chronic phase, accelerated disease or after treatment for blast crisis or RAEB or RAEBT stages of MDS which have not responded to or recurred following induction therapy. Furthermore, the patient's leukemic or MDS blasts should be documented to express the WT1 protein detectable by immunohistopathologic analysis of diagnostic paraffin embedded marrow biopsies, obtained at diagnosis of relapse or be of a type known to commonly express WT1 at high frequency. Expression of WT1 will be assessed by a modification of the technique of Dupont and Soslow (36) and graded according to an adaptation of the German Immunoreactive Score (IRS) which is the product of subscores for intensity of immunoreactivity (0-3+) and distribution of immunoreactivity (0-4+). For this study, leukemic blasts with IRS scores of 4-12 will be considered positive.
* A pathologically confirmed diagnosis of leukemia or MDS.
* Patients who have already received an allogeneic hematopoietic cell transplant and have either a documented relapse of leukemia or MDS or have recurrent persistent minimal residual disease as documented by at least 2 sequential testings, separated by 1 week, demonstrating molecular evidence of leukemia or MDS by FISH, cytogenetics or fluorescent immunocytometry.
* Patients who are to receive an allogeneic hematopoietic cell transplant as treatment for a leukemia or myelodysplastic syndrome that has an expected risk of relapse exceeding 30% will be eligible to have donor-derived WT1 peptide sensitized T cells generated prior to or at the time of transplant for immediate use post transplant at such time that the patient is found to have minimal residual disease or relapse. This includes patients with:
* ALL, AML or MDS refractory to primary induction therapy
* ALL or AML at any stage later than 1° relapse
* CML in 2° or greater chronic phase after chemotherapy
* CML in persistent accelerated phase or blast crisis
* High risk MDS (RAEB and RAEB+) which has failed to respond or has recurred following induction chemotherapy
* The patients' leukemia or MDS blasts must express the WT1 protein detectable by immunohistopathologic analysis, or; if an adequate sample is not available for testing, , must have a form of leukemia (ALL, AMLs other than M5) or MDS (2° MDS, RAEB, RAEBT) known to over express WT1 in a high proportion of cases (>60%). For patients who develop a documented relapse of leukemia or MDS following transplant, marrow aspirates should be evaluated for the proportion of blasts expressing WT1 by immunohistology or FACS whenever possible.
* The patient's hematopoietic cell transplant donor must consent to a 2 volume leukapheresis or whole blood donations obtained at one phlebotomy which, will total approximately 250 ml from which the WT-1 specific T cells to be used for adoptive transfer will be generated
* KPS or Lansky score > or equal to 40
* Adequate bone marrow, renal and hepatic function at the time of treatment with WT1 specific T cells:
* Absolute neutrophil count (ANC) > or equal to 1000/mm3, with or without G-CSF support.

This requirement may be waived if the patient has hematologic relapse of disease or if patient has not yet recovered counts from chemotherapy.

* Platelets > or equal to 20,000/mm3. This requirement may be waived if patient has hematologic relapse of disease or if patient has not yet recovered counts from chemotherapy.
* Creatinine < than or equal to 2.0mg/dL
* ALT, AST <3.0 and total bilirubin all < 2.5 x the institutional ULN
* There are no age restrictions to this protocol.
* Patients with relapse also detected in the CNS may be treated on this protocol. However, if intrathecal chemotherapy is being administered, T cells should not be administered until at least 24 hours thereafter.

Exclusion Criteria:

* Patients with active (grade 2-4) acute graft vs. host disease (GVHD), chronic GVHD or an overt autoimmune disease (e.g. hemolytic anemia) requiring high doses of glucocorticosteroid (>0.5 mg/kg/day prednisone or its equivalent) as treatment.
* Patients with other conditions not related to leukemic relapse (e.g. veno-occlusive disease or uncontrolled bacterial, viral or invasive fungal infection) which are also life-threatening and which would preclude evaluation of the effects of a T cell infusion.
* Patients who are pregnant.

Donor Eligibility for Donation of Blood Lymphocytes for Generation of Donor-Derived WT-1-Specific T Cells.

The eligibility criteria for the donor of blood to be used to generate WT1 peptide sensitized T cells are:

* The donor of WT-1 specific T. lymphocytes will be the same donor who provided the patient's hematopoietic stem cell transplant (HSCT). These normal donors will be evaluated for evidence of prior sensitization to EBV by EBV serology. If the donor is seropositive, and donor T cells are sensitized with the donor's WT-1 peptide- loaded EBV transformed B cells, EBV-specific T-cells will also be generated from seropositive donors generating WT-1 specific T-cells, and their growth and persistence post transfer will be compared to that of the WT 1 specific T-cells.
* Since the donor will have already undergone an extensive evaluation of his/her health to ascertain eligibility for donating the patient's HSCT, re-evaluation for this blood donation will be limited to a clinical history, physical examination and blood tests to insure against any new condition which, in the opinion of the donor's physician, preclude the donor from donating the blood required.
* New health conditions which would exclude a transplant donor from a second blood donation are limited, but include:
* New onset of an HIV infection
* Other uncontrolled infection which could be transmitted to the patient by blood cells and would place the patient at significant increased risk of severe morbidity or death.
* Significant anemia with Hgb < than or equal to 10 gm/dl, persisting since the time of the original transplant donation.
* History of myocardial infarction or stroke since the time of HSCT donation which might increase the risk of blood donation. A perspective donor will be informed of the purposes of this study, and its requirements. If he/she consents, the donor will be requested to provide two blood samplings.
* An initial donation of 25ml blood anticoagulated with heparin or ACD. This blood is used to establish a B cell line transfused transformed with the B95.8 laboratory strains of EBV. This EBV+ B cell line/ (EBVBLCL) will be used as an antigen-presenting cell. When loaded with the pool of WT-1 pentadecapeptides, the EBVBLCL efficiently sensitize T cells from the same donors against WT-1 as well as EBV.

Because the establishment and testing of an EBV transformed B cell line suitable for use as an antigen-presenting cell require 4-5 weeks of in vitro culture, it is important that this sample be obtained as early as possible for patients at risk for leukemic relapse, since disease relapse most frequently occurs 2-6 months post transplant. Accordingly, this blood sample should be obtained from the donor prior to donation of the hematopoietic progenitor cell transplant whenever possible.

* A donation of either a single standard 2 blood volume leukapheresis collected in standard ACD anticoagulant. If it is impossible to collect a leukapheresis from some of the donors, a unit of whole blood will be accepted by the AICTF (Adoptive Immune Cell Therapy Facility manufacturing the clinical grade cell products under GMP conditions in MSKCC) for the generation of limited number of T cells. This blood is required for isolation of the T cells to be sensitized with the pool of WT-1 15-mers loaded on autologous dendritic cells or autologous EBVBLCL, and propagated in vitro. In addition, it is required to provide autologous feeder cells essential to sustain T-cell growth without the risk of stimulating the growth of alloreactive T-cells capable of inducing GVHD.
* This donation of a leukapheresis or a unit of blood will be obtained from unrelated HSCT donors at least 2 weeks after their donation of an HSCT, but soon thereafter as possible.

In addition to providing written consent to these donations of blood for the purpose of generating WT-1-specific T-cells for potential use in the treatment of recurrent leukemia or persistent residual disease developing in the patient for whom the donor has provided an HSCT, each donor will be informed of and asked to provide separate consent to each of the following potential applications of the blood cells donated:

* The use of a fraction of the cells isolated to generate immune T-cells specific for viruses, such as Epstein-Barr virus (EBV) and cytomegalovirus (CMV) ,that can cause lethal infections or lymphomas in transplant recipients. Such T-cells could then be used, under separate protocols, to treat EBV-associated diseases (IRB 95-024) and/or to treat CMV infections (IRB 05-065) in the patient receiving the donor's hematopoietic progenitor cell transplant.

Consenting to this application will limit the number of blood donations that would be required of any donor, since the white cells donated in a leukapheresis should provide enough cells to grow immune T-cells against WT-1, EBV and CMV.

The donation of immune T-cells specific for EBV or CMV generated from the donor that are not used for or required by the patient for whom they were originally intended to a bank of immune cells that will be started and maintained cryopreserved under GMP conditions in the Adoptive Immune Cell Therapy Facility at MSKCC, for potential use in the treatment of other patients with EBV lymphomas or cytomegalovirus infections that express HLA alleles shared by the donor.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-02-08 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
assess toxicity of in vitro expanded allogeneic WT1 peptide-specific T-cells derived from transplant donor,when given to patients with leukemia or other WT1+ hematologic malignancy having relapsed after transplant or persistent minimal residual disease | conclusion of the study

SECONDARY OUTCOMES:
to assess the effects of the adoptively transferred T cells on the progression of disease | conclusion of the study
to quantitate the number of WT1 peptide-specific T cells in the blood at defined intervals post infusion in order to determine their survival and proliferation in the host. | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Susan Prockop, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org